CLINICAL TRIAL: NCT03628872
Title: Treatment of Periodontitis Utilizing Two Different Modalities: Erbium-doped Yttrium Aluminium Garnet (Er:YAG) Laser and Conventional Mechanical Debridement
Brief Title: Treatment of Periodontitis With Er:YAG Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Philip Y. Kang, Assistant Professor of Dental Medicine (Periodontist) at the Columbia University Medical Center, College of Dental Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR6077
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Generalized Moderate Chronic Periodontitis; Generalized Severe Chronic Periodontitis; Periodontal Diseases
Keywords: Scaling and root planing; Laser scaling
MeSH Terms: conditions — Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Examiner was blinded to treatment allocation during baseline and at the 3 month re-evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scaling and Root Planing with Hand Instruments (Active Comparator): Patients will undergo scaling and root planing with hand instruments (half of their mouth, following a split-mouth design)
  Interventions: Procedure: Scaling and root planing; Device: Hand instruments
- Er:YAG Laser Scaling (Experimental): Patients will undergo scaling and root planing with Er:YAG Laser in the untreated half of their mouth.
  Interventions: Procedure: Scaling and root planing; Device: Er:YAG Laser

INTERVENTIONS:
Procedure: Scaling and root planing — A non-surgical procedure that treats periodontal disease, sometimes called a deep cleaning, is considered the "gold standard" (standard of care) of treatment for patients with chronic periodontitis.
  Other Names: Deep cleaning
Device: Er:YAG Laser — This laser is intended to be used for dental surgery. The Er:YAG Laser emits an infrared beam which is readily absorbed by water contained by both hard and soft tissues of the human body. As a result, energy of the laser beam instantly vaporizes the water molecules in soft and hard tissues of the tooth and surrounding tissues causing the tissues to crumble away or resection of the soft tissues of gingival.
  Other Names: Erbium-doped Yttrium Aluminium Garnet Laser
  Arms: Er:YAG Laser Scaling
Device: Hand instruments — 11/12 and 13/14 gracey, 4R/4L curette and sickle - standard of care choices for performing scaling and root planing.
  Other Names: Hand instrumentation
  Arms: Scaling and Root Planing with Hand Instruments

SUMMARY:
The purpose of this research project is to gain information on the best and most comfortable way to treat the periodontal disease. The main objective is to compare the efficacy of conventional scaling and root planning compared to laser scaling for the non-surgical treatment of periodontal disease. Both therapies have shown to be effective and are regularly used in the dental clinic.

DETAILED DESCRIPTION:
The study has been designed as a single blinded split-mouth randomized controlled clinical trial. Patients will be randomized prior to treatment, to which the examiner will be blinded. Clinical parameters will be recorded at baseline and 3 months after treatment has been completed. At the time of recruitment, inclusion/exclusion criteria checklist, informed consent and baseline measurements will be obtained and recorded. Medical history will be updated and radiographs will be reviewed or taken. During the second appointment, conventional scaling and root planing will be performed in the corresponding quadrant; during the third appointment, laser therapy will be conducted, 1 month after, during the forth appointment, a follow up (no measurements) will be scheduled with provider, and 3 months after scaling completion, measurements will be taken and periodontal maintenance performed. Patient will receive home care instructions at every visit and will fill out a visual analogue scale at baseline, 1 month and 3 month visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Informed Consent
* Good general health
* Participants > 18 years of age
* Participants with > 20 teeth with 5 teeth, including at least 1 molar, in each quadrant of the mouth
* Participants with > 30% of the present teeth with Probing depths of > 4mm and Bleeding on Probing
* Non-smoker and former smokers (stopped smoking > 1 year)
* Participants that have not received any periodontal treatment in the past 3 months

Exclusion Criteria:

* Participants with uncontrolled systemic diseases that could affect the treatment outcome such as Diabetes with HbA1c > 7.0 percent, rheumatoid arthritis, immunosuppression, HIV with detectable viral loads
* Participants requiring antibiotic prophylaxis for any cardiovascular conditions or after any transplant and/or replacement procedures
* Pregnant women
* Patients treated with systemic antibiotic therapy of periodontal/mechanical/local delivery therapy within 6 weeks prior to study entry and throughout the study duration
* Patients being chronically (two weeks or more) treated with any NSAIDs, steroids or any medications known to affect soft tissue condition (excluding treatment with Acetylsalicylic acid < 100 mg/day)
* Presence of orthodontic appliances, or any removable appliances that impinges on the tissues being assessed.
* Presence of soft or hard tissue tumors of the oral cavity
* The presence of any medical or psychiatric condition or any other condition that, in the opinion of the Investigator, could affect the successful participation of the patient in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kang, DDS, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Dental Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The same 26 patients received both interventions. Each patient's right and left sides (mouth quadrants) were randomly assigned to receive one of the two treatment modalities using random sequences generated by a software application: conventional scaling and root planing (C-SRP), or conventional scaling with Er:YAG laser-assisted scaling and root planing (L-SRP).
Units Other Than Participants: mouth quadrant
Groups:
- Conventional Scaling and Root Planing: Conventional Scaling and Root Planing with hand instruments were randomly assigned to the left or the right mandible side in a split-mouth randomized design.
  Scaling and root planing: A non-surgical procedure that treats periodontal disease, sometimes called a deep cleaning, is considered the "gold standard" (standard of care) of treatment for patients with chronic periodontitis.
  Hand instruments: 11/12 and 13/14 gracey's, mini 11/12 and 13/14 gracey's, 4R/4L curette and sickle scaler - the standard of care choices for performing scaling and root planing.
- Er:YAG: Conventional Scaling and Root Planing with Er:YAG laser were randomly assigned to the left or the right mandible side in a split-mouth randomized design.
  Er:YAG Laser: This laser is intended to be used for dental surgery. The Er:YAG laser emits an infrared beam which is readily absorbed by water contained by both hard and soft tissues of the human body. As a result, energy of the laser beam instantly vaporizes the water molecules in soft and hard tissues of the tooth and surrounding tissues causing the tissues to crumble away or resection of the soft tissues of gingival.
Period: Overall Study
Arm/Group | Conventional Scaling and Root Planing | Er:YAG
Started | 26; 52 mouth quadrant | 26; 52 mouth quadrant
Completed | 26; 52 mouth quadrant | 26; 52 mouth quadrant
Not Completed | 0; 0 mouth quadrant | 0; 0 mouth quadrant

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Patients will undergo a split-mouth design, with one half side of the mouth (one side has 2 quadrants which include the upper and lower mouth) receiving non-surgical treatment with conventional scaling and root planing with hand instruments, and the other half side of their mouths receiving non-surgical treatment with conventional scaling and root planing with Er:YAG laser.
  Scaling and root planing: A non-surgical procedure that treats periodontal disease, sometimes called a deep cleaning, is considered the "gold standard" (standard of care) of treatment for patients with chronic periodontitis.
  Hand instruments: 11/12 and 13/14 gracey's, mini 11/12 and 13/14 gracey's, 4R/4L curette and sickle scaler - the standard of care choices for performing scaling and root planing.
  Er:YAG Laser: This laser is intended to be used for dental surgery. The Er:YAG laser emits an infrared beam which is readily absorbed by water contained by both hard and soft tissues of the human body. As a result, energy of the laser beam instantly vaporizes the water molecules in soft and hard tissues of the tooth and surrounding tissues causing the tissues to crumble away or resection of the soft tissues of gingival.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 52.21 [33 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  African American | 5
  Hispanic | 15
  Asian | 2
  Not reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment Level (CAL)
Description: Calculated based on distance from CEJ to gingival margin and the pocket depth (site specific measurement)
Time Frame: 3 months after treatment
Population: The same 26 patients participated in both arms, where half side of their mouths (52 quadrants - one side has two quadrants) were treated with conventional scaling and root planing and the other half side of their mouths (52 quadrants on the other side) were treated with Er:YAG laser.
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: Mouth quadrant
Groups:
- Conventional Scaling and Root Planing: Patients will undergo non-surgical treatment with conventional scaling and root planing with hand instruments or Er:YAG following a split-mouth design (both upper and lower quadrants on each side were treated).
  Scaling and root planing: A non-surgical procedure that treats periodontal disease, sometimes called a deep cleaning, is considered the "gold standard" (standard of care) of treatment for patients with chronic periodontitis.
  Hand instruments: 11/12 and 13/14 gracey's, mini 11/12 and 13/14 gracey's, 4R/4L curette and sickle scaler - the standard of care choices for performing scaling and root planing.
- Er:YAG: Patients will undergo non-surgical treatment with conventional scaling and root planing with hand instruments or Er:YAG following a split-mouth design (both upper and lower quadrants on each side were treated).
  Er:YAG Laser: This laser is intended to be used for dental surgery. The Er:YAG laser emits an infrared beam which is readily absorbed by water contained by both hard and soft tissues of the human body. As a result, energy of the laser beam instantly vaporizes the water molecules in soft and hard tissues of the tooth and surrounding tissues causing the tissues to crumble away or resection of the soft tissues of gingival.
Arm/Group | Conventional Scaling and Root Planing | Er:YAG
Number analyzed (Participants) | 26 | 26
Number analyzed (Mouth quadrant) | 52 | 52
mm | 3.5 (0.7) | 3.4 (0.4)

2. Primary Outcome: Change in Pocket Depth (PD)
Description: Measured at 6 sites per tooth in millimeters (mm) (site specific measurement). The mean value of the measurements was obtained for both treatment groups by averaging all teeth for each quadrant.
Time Frame: 3 months after treatment
Population: The same 26 patients participated in both arms, where half of their mouths (52 quadrants) were treated with conventional scaling and root planing and the other half of their mouths (52 quadrants) were treated with Er:YAG laser.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Mouth quadrant
Arm/Group | Conventional Scaling and Root Planing | Er:YAG
Number analyzed (Participants) | 26 | 26
Number analyzed (Mouth quadrant) | 52 | 52
mm | 3.12 (0.56) | 3.13 (0.49)

3. Secondary Outcome: Plaque Index (PI)
Description: Plaque and calculus accumulation on tooth surfaces (site specific measurement). Plaque Index is calculated by [number of sites with plaque] divided by [number of sites evaluated], multiplied by 100 (represented as a percent).
Time Frame: 3 months after treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: Mouth quadrant
Groups:
- Er:YAG Laser Scaling: Patients will undergo non-surgical treatment with conventional scaling and root planing with hand instruments or Er:YAG following a split-mouth design (both upper and lower quadrants on each side were treated).
  Er:YAG Laser: This laser is intended to be used for dental surgery. The Er:YAG laser emits an infrared beam which is readily absorbed by water contained by both hard and soft tissues of the human body. As a result, energy of the laser beam instantly vaporizes the water molecules in soft and hard tissues of the tooth and surrounding tissues causing the tissues to crumble away or resection of the soft tissues of gingival.
Arm/Group | Conventional Scaling and Root Planing | Er:YAG Laser Scaling
Number analyzed (Participants) | 26 | 26
Number analyzed (Mouth quadrant) | 52 | 52
percent | 61.16 (33.66) | 65.22 (32.21)

4. Secondary Outcome: Bleeding on Probing (BoP)
Description: Bleeding after probing the pocket (site specific measurement). BoP is calculated by: [number of bleeding sites] divided by [number of sites evaluated], multiplied by 100 (represented as a percent).
Time Frame: 3 months after treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Units Other Than Participants: Mouth quadrant
Arm/Group | Conventional Scaling and Root Planing | Er:YAG Laser Scaling
Number analyzed (Participants) | 26 | 26
Number analyzed (Mouth quadrant) | 52 | 52
percent | 29.21 (23.92) | 31.34 (22.22)

5. Secondary Outcome: Average Duration of Treatment
Description: Comparison of duration of treatment between the 2 modalities
Time Frame: Time between the start of treatment to treatment completion, up to 180 minutes
Population: as for outcome 2
Measure: Mean (Full Range); unit: minutes
Units Other Than Participants: Mouth quadrant
Arm/Group | Conventional Scaling and Root Planing | Er:YAG
Number analyzed (Participants) | 26 | 26
Number analyzed (Mouth quadrant) | 52 | 52
minutes | 92.04 [60 to 138] | 54.15 [40 to 82]

6. Secondary Outcome: Number of Participants Who Preferred Modality
Description: Participants were given 2 multiple choice questions to assess their modality of preference and the reasoning behind it.
Time Frame: 3 months after treatment
Measure: Number; unit: participants
Arm/Group | Conventional Scaling and Root Planing | Er:YAG
Number analyzed (Participants) | 26 | 26
participants
  Participants who preferred Er:YAG Laser modality | 21 | 21
  Participants who preferred Conventional Scaling and Root Planning modality | 0 | 0
  Participants who had no preference between the 2 modalities | 5 | 5

7. Secondary Outcome: Number of Patients Who Experienced a Better Improvement in Sensitivity
Description: A numeric scale was completed by participants to assess their degree of sensitivity or pain with a modified 0 - 10 scale (i.e.: 0- no pain/sensitivity; 5- moderate pain or sensitivity, may require medication; 10- unbearable sensitivity or pain that impairs my sleep). Baseline and 3 months reported scores were compared within each patient and between modalities. The numbers reported are participants that experienced a better improvement in sensitivity within the respective modality.
Time Frame: Baseline and 3 months
Population: 9 patients experienced no differences in sensitivity according to the modality.
Measure: Number; unit: participants
Arm/Group | Conventional Scaling and Root Planing | Er:YAG
Number analyzed (Participants) | 26 | 26
participants | 0 | 17

ADVERSE EVENTS:
Time Frame: 3 months after treatment.
Groups:
- Scaling and Root Planing With Hand Instruments: Adverse Events localized to the mouth side treated with hand instruments.
- Scaling and Root Planing With Er:YAG Laser: Adverse Events localized to the mouth side treated with Er:YAG Laser.
- All Participants: All Adverse Events, including those that affected participants as a whole (systemic events).
Arm/Group | Scaling and Root Planing With Hand Instruments | Scaling and Root Planing With Er:YAG Laser | All Participants
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT03628872/Prot_SAP_001.pdf